CLINICAL TRIAL: NCT06385483
Title: MATCH Treatment Subprotocol A: Phase II Trial of Afatinib in Patients With Solid Tumors (Other Than Small Cell and Non-Small Cell Lung Cancer) or Lymphomas, That Have Activating Mutations of EGFR and Have Progressed After Standard Treatment
Brief Title: Testing Afatinib as Potentially Targeted Treatment in Cancers With EGFR Genetic Changes (MATCH - Subprotocol A)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01125; NCI-2024-01125 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-A (Other: ECOG-ACRIN Cancer Research Group); EAY131-A (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-04-25; First posted 2024-04-26 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Afatinib; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Nuclear Medicine Department, Hospital

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (afatinib) (Experimental): Patients receive afatinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients may also undergo ECHO or nuclear study throughout the trial as clinically necessary. Patients undergo biopsies and blood sample collection on study.
  Interventions: Drug: Afatinib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Radionuclide Imaging

INTERVENTIONS:
Drug: Afatinib — Given PO
  Other Names: BIBW 2992; BIBW-2992; BIBW2992
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Radionuclide Imaging — Undergo nuclear study
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy

SUMMARY:
This phase II MATCH treatment trial tests how well afatinib works in treating patients with cancer that has certain genetic changes. Afatinib is in a class of medications called kinase inhibitors. It is used in patients whose cancer has a certain mutation (change) in the EGFR gene. It works by blocking the action of mutated EGFR that signals cancer cells to multiply. This helps to stop or slow the spread of cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive afatinib orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and on study, as well as during follow-up as clinically necessary. Patients also undergo echocardiography (ECHO) or nuclear study throughout the trial as clinically necessary. Patients undergo biopsies and blood sample collection on study.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must fulfill all eligibility criteria of MATCH Master Protocol at the time of registration to treatment step (Step 1, 3, 5, 7)
* Patient's tumor must have either of the below, or another aberration, as determined via the MATCH Master Protocol:

  * Activating mutations of EGFR (del 19, L858R) OR
  * Any malignancy harboring any of the following mutations: EGFR G719A, G719C, G719D, G719S EGFR L861Q, EGFR S768I
  * Tumors with an exon 20 insertion alone without the above mutations will be excluded, with the exception of exon 20 insertions approved as inclusion variants as part of the dynamic actionable mutation of interest (aMOI) process
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients with known left ventricular dysfunction must have ECHO or a nuclear study (multigated acquisition scan [MUGA] or first pass) within 4 weeks prior to registration to treatment and must not have left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible

  * NOTE: Pre-treatment LVEF determination in patients without known left ventricular dysfunction is NOT otherwise required
* Patients must not have known hypersensitivity to afatinib or compounds of similar chemical or biologic composition
* Patients must have =< grade 1 renal function as defined below:

  * Creatinine =< 1.5 x normal institutional limits OR
  * Measured creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal or as calculated by the Cockcroft-Gault equation
  * The above renal eligibility criteria should be strictly followed and will override the MATCH Master Protocol requirements
* Patients must not have had prior treatment with an EGFR tyrosine kinase inhibitor (TKI) (e.g. afatinib, erlotinib, gefitinib, neratinib, dacomitinib, AZD9291, cabertinib, CO-1686)
* Patients with non-small cell lung cancer and small cell lung cancer will be excluded
* Patients with a history of interstitial lung disease will be excluded
* Patients with glioblastoma multiforme (GBM) will be excluded
* Patients must have =< grade 1 diarrhea at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Scott N Gettinger, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol A was activated on August 12, 2015. Nineteen patients were enrolled between February 2018 and January 2020. All patients were enrolled though the outside laboratory and had their samples centrally confirmed.
Pre-assignment Details: EGFR variants allowing entry into subprotocol A included classic activating deletion 19 and L858R EGFR mutations, EGFR G719A, G719C, G719D, G719S, L861Q, and S768I. The mutation status was determined by a CLIA-approved assay performed in an NCI-MATCH approved laboratory, these cases had to be confirmed to be used in primary analysis.
Groups:
- Treatment (Afatinib): Patients receive afatinib 40 mg PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients may also undergo ECHO or nuclear study throughout the trial as clinically necessary. Patients undergo biopsies and blood sample collection on study.
Period: Overall Study
Arm/Group | Treatment (Afatinib)
Started | 19
Started Protocol Therapy | 17
Eligible, Treated and Mutation Status Confirmed (Primary efficacy analysis set) | 17
Completed | 0
Not Completed | 19
Not completed — Withdrawal by Subject | 2
Not completed — Never start protocol therapy | 2
Not completed — Disease progression | 15

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 58 [41 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 17
percentage of participants | 11.8 [2.1 to 32.6]

2. Secondary Outcome: 6-month Progression Free Survival (PFS)
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 17
percentage of participants | 15 [0 to 30.7]

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 17
months | 1.7 [1.35 to 1.94]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Seventeen patients were included in the toxicity analysis (excluding two who did not receive treatment).
Arm/Group | Treatment (Afatinib)
All-Cause Mortality (participants affected / at risk) | 16/19
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Afatinib) (N=17)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Afatinib) (N=17)
Anemia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 12
Dysphagia (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Paronychia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT06385483/Prot_000.pdf